CLINICAL TRIAL: NCT05819281
Title: Efficacy of a Probiotic Blend to Reduce Gastrointestinal Symptoms and Improve Quality of Life in Patients Diagnosed With Irritable Bowel Syndrome
Brief Title: Efficacy of a Probiotic Blend to Reduce Gastrointestinal Symptoms in Patients With Irritable Bowel Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Responsible Party: Principal Investigator, Monique Michels, Principal Investigator, Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 63067022.2.0000.0119
Record Dates: First submitted 2023-02-09; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic blend group (Experimental): Volunteers supplemented with the probiotic product (n=57) (Lactobacillus acidophilus, Lactobacillus paracasei, Bifidobacterium lactis, Bifidobacterium bifidum e Lactobacillus rhamnosus - Final concentration: 1 x 10e10 CFU/day).
  Interventions: Dietary Supplement: Probiotic blend
- Placebo group (Placebo Comparator): Placebo Group (n=57): Volunteers supplemented with placebo (maltodextrin)
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: Probiotic blend — (Lactobacillus acidophilus, Lactobacillus paracasei, Bifidobacterium lactis, Bifidobacterium bifidum e Lactobacillus rhamnosus - Final concentration: 1 x 1010 CFU/day).
  Arms: Probiotic blend group
Dietary Supplement: PLACEBO — Maltodextrin
  Arms: Placebo group

SUMMARY:
Irritable bowel syndrome (IBS) is a recurrent, functional disorder characterized by abdominal pain and discomfort, changes in bowel habits and gastrointestinal symptoms such as distension and sensation of abdominal inflammation, incomplete evacuation, urgency and tenesmus. In addition to gastrointestinal symptoms, patients with IBS often experience a wide range of other problems, such as non-abdominal pain, psychological symptoms, poor quality of life, and difficulties in carrying out activities of daily living. Studies carried out with probiotics have shown that their administration can be effective in the prevention and treatment of IBS. Our objective is to develop a probiotic product (Lactobacillus acidophilus, Lactobacillus paracasei, Bifidobacterium lactis, Bifidobacterium bifidum e Lactobacillus rhamnosus) is safe and effective in reducing symptoms caused by IBS, as well as improving quality of life. In the present study, 114 volunteers of both genders will be included, randomly distributed into two groups: Test group (n=57): Volunteers supplemented with the probiotic product (Lactobacillus acidophilus, Lactobacillus paracasei, Bifidobacterium lactis, Bifidobacterium bifidum e Lactobacillus rhamnosus- Final concentration: 1 x 1010 CFU/day). Placebo Group (n=57): Volunteers supplemented with placebo. The study will last 90 days and will have 3 visits to apply the proposed questionnaires.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a recurrent, functional disorder characterized by abdominal pain and discomfort, changes in bowel habits and gastrointestinal symptoms such as distension and sensation of abdominal inflammation, incomplete evacuation, urgency and tenesmus. This disorder affects men and women of all age groups, with a worldwide prevalence of 10% to 20%. In addition to gastrointestinal symptoms, patients with IBS often experience a wide range of other problems, such as non-abdominal pain, psychological symptoms, poor quality of life, and difficulties in carrying out activities of daily living. Treatment is usually symptomatic and associated with changes in lifestyle and diet, drug and psychological treatments and the use of probiotics. Studies carried out with probiotics have shown that their administration can be effective in the prevention and treatment of IBS. Furthermore, certain compositions of specific probiotics are found to have benefits, especially in quality of life, bloating and abdominal pain.

The hypothesis is that the use of a probiotic blend can reduce gastrointestinal symptoms and improve quality of life through its immunomodulatory and intestinal regulation mechanisms in patients with IBS

aim: To develop a safe and effective probiotic product (Lactobacillus acidophilus, Lactobacillus paracasei, Bifidobacterium lactis, Bifidobacterium bifidum e Lactobacillus rhamnosus) to reduce the symptoms caused by IBS.

METHODS

Randomized, double-blind, placebo-controlled study to evaluate the effectiveness of a probiotic blend (Lactobacillus acidophilus, Lactobacillus paracasei, Bifidobacterium lactis, Bifidobacterium bifidum e Lactobacillus rhamnosus) in improving symptoms caused by Bowel Syndrome Irritable (IBS). Study will be conducted with patients diagnosed with IBS by the gastroenterologist participating in the study, being an adult audience (18 - 65 years old). In the present study, 114 volunteers of both sexes will be included, randomly distributed into two groups:

Test group (n=57): Volunteers supplemented with the probiotic product (Lactobacillus acidophilus, Lactobacillus paracasei, Bifidobacterium lactis, Bifidobacterium bifidum e Lactobacillus rhamnosus - Final concentration: 1 x 1010 CFU/day). Placebo Group (n=57): Volunteers supplemented with placebo. The study will last for 90 days.

During the trial period, participants must attend the Research Center for the following visits:

Visit 1 (day 0) - Evaluation of inclusion and exclusion criteria, clinical and physical evaluation, presentation of the research and signing of the Free and Informed Consent Form in writing, partial delivery of the test product or placebo, delivery and application of questionnaires (questionnaires quality of life (by the SF-36 scale); Bristol scale, Gastrointestinal Symptom Rating Scale (GSRS) questionnaire for gastrointestinal evaluation and mental health questionnaire (BDI and IDATE questionnaire). The questionnaires will be applied preferably in person by the researchers involved (with scheduled time) in interview format or online via Google Forms form, providing confidentiality to all information collected. In addition, the first visit also An explanation will be given regarding the importance of the questionnaires, correct completion, and possible changes in the TGI in the first days of using the probiotic.

Visit 2 (day 45) - Clinical consultation with a specialist physician, final delivery of the test product or placebo, and application of questionnaires.

Visit 3 (day 90) - Clinical consultation with a specialist physician and final application of questionnaires. Closure of the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of Free and Informed Consent in writing, signed and dated;
* Age according to the indicated population;
* Patients diagnosed with IBS by a specialist.

Exclusion Criteria:

* Individuals with a history of daily consumption of probiotics, fermented milk and / or yogurt; subjects known to have demonstrated a prior reaction, including anaphylaxis, to any substance in the composition of the study product;
* Individuals who have unbalanced blood pressure; hx of heart disease, including valvulopathies or any implantable device; individuals on immunosuppressive therapy or any health condition causing immunosuppression; individuals with active, uncontrolled bowel disease such as Crohn's disease or ulcerative colitis;
* Women who are pregnant at the time of enrollment or who plan to become pregnant during the study;
* Individuals with concomitant participation in another clinical trial;
* History of autoimmune disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Bristol scale | Three times (0, 45 and 90 days after inclusion)
  The Bristol Stool Form Scale is used for describing feces into seven categories. Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 indicating lack of dietary fiber, and 6 and 7 indicate diarrhoea. People with irritable bowel syndrome (IBS) typically report that they suffer with abdominal cramps and constipation. In some patients, chronic constipation is interspersed with brief episodes of diarrhoea; while a minority of patients with IBS have only diarrhoea.

SECONDARY OUTCOMES:
Change of quality of life (SF-36 scale) | Three times (0, 45 and 90 days after inclusion)
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study for the objective measure of the quality of life. The SF-36 includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions.
  It comprises 36 questions that cover eight domains of health
Change of mental health - depression | Three times (0, 45 and 90 days after inclusion)
  The Beck Depression Scale or Beck Depression Inventory (BDI, BDI-II), consists of a self-report questionnaire with 21 multiple-choice items. It is one of the most used instruments to measure the severity of depressive episodes. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Gastrointestinal Symptom Rating Scale (GSRS) | Three times (0, 45 and 90 days after inclusion)
  The GSRS is a disease-specific instrument. The 15 items combine into five symptom clusters: Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The reliability and validity of the GSRS are well-documented, and norm values for a general population are available. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Change of mental health - anxiety | Three times (0, 45 and 90 days after inclusion)
  The State-Trait Anxiety Inventory (STAI) is one of the most used instruments to quantify subjective components related to anxiety. It consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety and trait anxiety. Higher scores are positively correlated with higher levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Do Extremo Sul Catarinense, Criciúma, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol